CLINICAL TRIAL: NCT00730340
Title: Decreased Morbidity With Closure of the Tonsillar Fossae
Brief Title: Closure Method Study Following Tonsillectomy in Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Wayne E. Berryhill, M.D., University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tonsillar Closure_Berryhill
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Tonsillectomy; Children
Keywords: Tonsillectomy, tonsillar fossa, wound closure
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will receive closure of the tonsillar fossae following tonsillectomy.
  Interventions: Procedure: Closure of the Tonsillar Fossa
- 2 (Active Comparator): Patients will not receive closure to one or both tonsillar fossa following a tonsillectomy
  Interventions: Procedure: Tonsillectomy with open fossa

INTERVENTIONS:
Procedure: Closure of the Tonsillar Fossa — We hypothesize that closure of the tonsillar fossa decreases the morbidity of pain by decreasing exposure of the raw operative bed to oral secretions, mediation, and oral intake, and decreases the morbidity of post-operative hemorrhage by having the operative wound closed.
  Arms: 1
Procedure: Tonsillectomy with open fossa — SOP for a tonsillectomy.
  Arms: 2

SUMMARY:
This is a children's study evaluating the effects of a tonsillectomy with tonsillar fossae closure compared to without closure of the operative wound.

DETAILED DESCRIPTION:
This is a children's study. Patients experience significant postoperative pain, activity limitation and sometimes other significant postoperative complications. We are going to compare the effects of closing the tonsil wound versus non-closure. A daily journal will be kept (by the patient's parent or legal guardian)to log in measures of morbidity. Postoperative telephone calls will be made and scripted questions will be asked regarding any tonsillar hemorrhage requiring medical re-evaluation, and dehydration requiring medical re-evaluation. The patients will also be examined in the clinic at 10-14 days postoperatively to determine if the fossa remained closed or dehisced.

ELIGIBILITY:
Inclusion Criteria:

* Normal children between that ages of five to ten requiring a tonsillectomy

Exclusion Criteria:

* Children older than ten years of age.
* Those children with identified syndromes, cleft palates and velopharyngeal insufficiency will not be eligible.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Decreased morbidity in children with closure of the tonsillar fossae compared with tonsillectomy without closure | 6 months

SECONDARY OUTCOMES:
The patients will also be examined in the clinic postoperatively to determine if the fossae remained closed or dehisced. | 10-14 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wayne E Berryhill, M.D., Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States